CLINICAL TRIAL: NCT05032989
Title: Extraction of Distoangular and Vertically Positioned Mandibular 3rd Molars, A Comparative Study: Conventional Surgical Technique vs. Cowhorn Forceps Technique
Brief Title: Extraction of Distoangular and Vertically Positioned Mandibular 3rd Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Syed Wajid Hasan, Postgraduate Trainee, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: wajid001
Record Dates: First submitted 2021-08-31; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extraction of distoangular and vertically positioned 3rd molar using cowhorn forcep (Experimental): Extraction with new technique
  Interventions: Procedure: Extraction of mandibular 3rd molar via Cowhorn forcep technique
- Extraction of distoangular and vertically positioned 3rd molar via conventional method (Active Comparator): Extraction with the conventional technique
  Interventions: Procedure: Extraction of mandibular 3rd molar via conventional technique

INTERVENTIONS:
Procedure: Extraction of mandibular 3rd molar via Cowhorn forcep technique — Cowhorn forceps technique used to extract the tooth results in less post operative pain and swelling also it makes the extraction easier.
  Arms: Extraction of distoangular and vertically positioned 3rd molar using cowhorn forcep
Procedure: Extraction of mandibular 3rd molar via conventional technique — Conventional method of extraction uses dental elevator and forceps resulting in post operative pain and swellig.
  Arms: Extraction of distoangular and vertically positioned 3rd molar via conventional method

SUMMARY:
Mandibular 3rd molars are the most commonly impacted teeth in oral cavity followed by maxillary 3rd molars and maxillary canines respectively. Impaction is a condition where a tooth fails to erupt in its final functional position, theoretically owing to inadequate space distal to the second mandibular molar and the anterior border of the ascending ramus of the mandible . Surgical removal of the third molar is the most common procedure carried out by a maxillofacial surgeon in the dental office. Surgical extractions are time consuming, expensive and cause morbidities such as pain, swelling, dry socket, trismus, and nerve injury when compared to non-surgical extractions. Various classifications have been proposed for mandibular 3rd molars, most common of which, is based on angulation of impacted tooth to the long axis of 2nd molar. Distoangular impacted 3rd molars are very difficult to remove because of lack of space distal to the tooth and lack of interdental space available for the application of elevator. Cowhorn forcep engages between the bifurcation of the mandibular molars and below the bone crest and causes displacement of tooth by upward movement or by splitting mesial and distal root. In our study cowhorn forcep are fist placed between 2nd and 3rd molar below the cementoenamel junction after its placement an apical pressure in applied and this rotation results an upward and distal movement and displacement of impacted tooth from the socket which then can easily be removed with cow horn forcep or molar crown forcep. The aim of our study is to present the minimal invasive technique for the extraction of distoangular and vertical impacted mandibular 3rd molars using cow horn forcep in comparison to conventional surgical techniques to avoid complications associated with open surgical techniques .

METHOD:

Total 128 patients will be recruited and divided into 64 patients in each group (two groups) attending in Dr. inshrat ul ebad institute of oral health sciences, Ojha, fulfilling inclusion criteria and undergoing extraction of 3rd molars will be included in this study. The participant will be briefed about the nature and purpose of the study. They will be ensured that their information will be used for the study purpose only. Informed consent from the participants will be obtained. Complete history from the patients will be taken and pre-operative evaluation will be done by clinical (pain and swelling) and radiographical (angulation of the tooth) examination. All the patients would undergo extraction of 3rd molars via both either conventional surgical technique or the proposed technique in the study. Followup will be done after 3 days to evaluate the same post-operative variables (pain and swelling) after extraction of 3rd molar and both techniques will then be compared in terms of variables measured.

DETAILED DESCRIPTION:
Mandibular 3rd molars are the most commonly impacted teeth in oral cavity followed by maxillary 3rd molars and maxillary canines respectively. Impaction is a condition where a tooth fails to erupt in its final functional position, theoretically owing to inadequate space distal to the second mandibular molar and the anterior border of the ascending ramus of the mandible . Surgical removal of the third molar is the most common procedure carried out by a maxillofacial surgeon in the dental office. Surgical extractions are time consuming, expensive and cause morbidities such as pain, swelling, dry socket, trismus, and nerve injury when compared to non-surgical extractions. Various classifications have been proposed for mandibular 3rd molars, most common of which, is based on angulation of impacted tooth to the long axis of 2nd molar. Distoangular impacted 3rd molars are very difficult to remove because of lack of space distal to the tooth and lack of interdental space available for the application of elevator. Cowhorn forcep engages between the bifurcation of the mandibular molars and below the bone crest and causes displacement of tooth by upward movement or by splitting mesial and distal root. In our study cowhorn forcep are fist placed between 2nd and 3rd molar below the cementoenamel junction after its placement an apical pressure in applied and this rotation results an upward and distal movement and displacement of impacted tooth from the socket which then can easily be removed with cow horn forcep or molar crown forcep.The aim of our study is to present the minimal invasive technique for the extraction of distoangular and vertical impacted mandibular 3rd molars using cow horn forcep in comparison to conventional surgical techniques to avoid complications associated with open surgical techniques .

Objective:

To compare the effectiveness of new technique using cow horn forcep with conventional surgical method among patients with vertical and distoangular lower third molar impactions requiring extraction.

Method:

Total 128 patients will be recruited and divided into 64 patients in each group (two groups) attending in Dr. inshrat ul ebad institute of oral health sciences, Ojha, fulfilling inclusion criteria and undergoing extraction of 3rd molars will be included in this study. The participant will be briefed about the nature and purpose of the study. They will be ensured that their information will be used for the study purpose only. Informed consent from the participants will be obtained. Complete history from the patients will be taken and pre-operative evaluation will be done by clinical (pain and swelling) and radiographical (angulation of the tooth) examination. All the patients would undergo extraction of 3rd molars via both either conventional surgical technique or the proposed technique in the study. Followup will be done after 3 days to evaluate the same post-operative variables (pain and swelling) after extraction of 3rd molar and both techniques will then be compared in terms of variables measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral distoangular and vertically positioned 3rd mandibular molars requiring extractions
* Bilateral partially impacted or erupted mandibular 3rd molars
* Both male and female patients
* Teeth which can be extracted by Intra-alveolar method under local anaesthesia
* Ages 18-35years

Exclusion Criteria:

* Patients refusing to sign the informed consent
* Patients that are medically compromised (systemic diseases)
* Teeth having radiographically evident large periapical changes (abscess/granuloma/cyst)
* Patients previously treated with radiotherapy or chemotherapy or both
* Carious mandibular 2nd molar or missing 1st molar

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Decrease post operative pain and swelling | 3rd post operative day
  cownhorn forcep technique is used to reduce post operative pain and swelling

CONTACTS AND LOCATIONS:
Overall Officials: Syed Wajid Hasan, BDS, Principal Investigator — DUHS